CLINICAL TRIAL: NCT05571033
Title: Operant Conditioning of the Soleus Stretch Reflex in Adults With Cerebral Palsy
Acronym: SRC-CP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burke Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRC-CP
Record Dates: First submitted 2022-10-02; First posted 2022-10-07 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Cerebral Palsy; Spastic Cerebral Palsy
Keywords: Hoffman Reflex; Spinal Reflex Conditioning
MeSH Terms: conditions — Cerebral Palsy; Reflex, Abnormal

STUDY DESIGN:
Intervention Model Description: Each participant will serve as their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinal reflex conditioning (Experimental): The OC intervention includes 6 baseline sessions and 24 conditioning/ no conditioning sessions held 3 times/week.
  To elicit an H-reflex, participants will be asked to stand in a comfortable position. Small pulses of energy will be applied to a nerve in the leg called the tibial nerve. We will record when the participant maintains leg muscle activity. During the intervention, participants will be trained to decrease their reflex in their calf.
  Interventions: Behavioral: Spinal reflex conditioning

INTERVENTIONS:
Behavioral: Spinal reflex conditioning — Each participant will serve as their own control. The intervention is 30 sessions. The first 6 sessions are baseline measures of reflexes. The remaining sessions will engage participants in learning how to decrease their reflex activity in their calf muscle on the more-affected leg. Each intervention visit will involve 20 trials in which participants do not get visual feedback about their performance, then 225 trials with visual feedback.

SUMMARY:
12 adults with spastic CP will complete 6 baseline sessions and 24 down conditioning sessions held 3 times/week. All clinical and physiological assessments collected at baseline will be reassessed after study completion, and follow ups after 2 weeks, 1 month and 3 months. The soleus H reflex (electric analogue of the stretch reflex) will be elicited in all sessions. In each session, participants will complete 20 baseline trials and 225 down conditioning trials to decrease the magnitude of the H-Reflex.

DETAILED DESCRIPTION:
Individuals with CP face significant challenges due to spasticity that causes activity and participation restrictions with increase in secondary conditions. This is caused by injury to the upper motor neurons causing disruption to the neural circuitry responsible for maintaining motor tone. A novel intervention, OC of the H reflex has shown promising effects to reduce spasticity and improve motor function in people with stroke and spinal cord. Its many known benefits include easy administration, non-invasive technique, no side effects, and long-term retention. In the study, the investigators will attempt to decrease the increased muscle tone of individuals with CP. If successful, it will not only provide evidence for future clinical application but also broaden the scope for alternate or supplementary non-invasive treatment approaches to decrease spasticity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above
2. Diagnosis of spastic Cerebral Palsy
3. Gross Motor Function Classification System level I-III
4. Stable medical background
5. Current medication will remain unchanged for 3 months
6. Provides informed consent
7. can walk at least 10 meters with or without assistive device
8. meets minimum study procedure requirements (elicitation of H-reflex).

Exclusion Criteria:

1. Pregnancy
2. uncontrolled diabetes
3. weak dorsiflexion
4. History of cardiac conditions
5. cognitive deficits that interfere with study procedure and steps for completion
6. Botox within 2 months of the study
7. H/O ankle surgeries in affected leg (Dorsal root rhizotomy etc.)
8. regular use of electrical stimulation to lower extremity muscles
9. Cochlear or metal implantations on body
10. No history of seizure after age 2 years
11. Current use of antiseizure medicines
12. Any metal or magnetic components in the head (surgical clips, metal work etc.)
13. Implanted device or cardiac pacemakers (applicable for DS8R too)
14. Skin disorders
15. Damaged skin (wounds, broken skin, or recent scar tissue)
16. Allergy to latex (tape)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Soleus H-Reflex size | Within one week before first intervention session to within one week after the end of intervention
  Size of h-reflex as measured by EMG
Attendance | At the end of the intervention, we will count the number of sessions each participant completed
  Measure of feasibility of protocol, whether or not people can attend all sessions

SECONDARY OUTCOMES:
10 meter walk test | Within one week before the first intervention session to within one week after the end of intervention
  Measure of how long it takes the participant to walk 10 meters
6 minute walk test | Within one week before the first intervention session to within one week after the end of intervention
  Measure the distance a participant can walk in 6 min
Fugl-Meyer | Within one week before the first intervention session to within one week after the end of intervention
  Standardized test of motor skill, range of motion, and spasticity
Modified Ashworth Scale | Within one week before the first intervention session to within one week after the end of intervention
  Measure of muscle spasticity in leg muscles
Range of motion | Within one week before the first intervention session to within one week after the end of intervention
  Measure of flexibility of leg joints
Fatigue Severity Scale | Within one week before the first intervention session to within one week after the end of intervention
  A survey of fatigue symptoms
Berg Balance Scale | Within one week before the first intervention session to within one week after the end of intervention
  Measure of participant's ability to balance
Timed up and Go | Within one week before the first intervention session to within one week after the end of intervention
  Measure of how quickly a participant can stand from a chair, walk, return to chair, and sit
Sit to Stand Test | Within one week before the first intervention session to within one week after the end of intervention
  Time it takes for a participant can stand up five times in a row
Patient Reported Outcome Measures (PROMIS) Anxiety question bank | Within one week before the first intervention session to within one week after the end of intervention
  computer-based survey for participants to answer questions about anxiety
Patient Reported Outcome Measures (PROMIS) Fatigue question bank | Within one week before the first intervention session to within one week after the end of intervention
  computer-based survey for participants to answer questions about fatigue
Patient Reported Outcome Measures (PROMIS) Depression question bank | Within one week before the first intervention session to within one week after the end of intervention
  computer-based survey for participants to answer questions about depression
Patient Reported Outcome Measures (PROMIS) General Life Satisfaction question bank | Within one week before the first intervention session to within one week after the end of intervention
  computer-based survey for participants to answer questions about General Life Satisfaction
Patient Reported Outcome Measures (PROMIS) General Self Efficacy question bank | Within one week before the first intervention session to within one week after the end of intervention
  computer-based survey for participants to answer questions about General Self Efficacy
Patient Reported Outcome Measures (PROMIS) Meaning and Purpose question bank | Within one week before the first intervention session to within one week after the end of intervention
  computer-based survey for participants to answer questions about Meaning and Purpose
Patient Reported Outcome Measures (PROMIS) Self-Efficacy for Managing Chronic Conditions question bank | Within one week before the first intervention session to within one week after the end of intervention
  computer-based survey for participants to answer questions about Self-Efficacy for Managing Chronic Conditions
Patient Reported Outcome Measures (PROMIS) Sleep Disturbances question bank | Within one week before the first intervention session to within one week after the end of intervention
  computer-based survey for participants to answer questions about sleep
Patient Reported Outcome Measures (PROMIS) Pain Interference question bank | Within one week before the first intervention session to within one week after the end of intervention
  computer-based survey for participants to answer questions about pain
Patient Reported Outcome Measures (PROMIS) Ability to Participate in Social Roles and Activities question bank | Within one week before the first intervention session to within one week after the end of intervention
  computer-based survey for participants to answer questions about Ability to Participate in Social Roles and Activities
Patient Reported Outcome Measures (PROMIS) Physical Function | Within one week before the first intervention session to within one week after the end of intervention
  computer-based survey for participants to answer questions about physical functioning
Patient Reported Outcome Measures (PROMIS) Satisfaction with Social Roles and Activities | Within one week before the first intervention session to within one week after the end of intervention
  computer-based survey for participants to answer questions about Satisfaction with Social Roles and Activities
Patient Reported Outcome Measures (PROMIS) Mobility question bank | Within one week before the first intervention session to within one week after the end of intervention
  computer-based survey for participants to answer questions about mobility
Patient Reported Outcome Measures (PROMIS) Social Isolation question bank | Within one week before the first intervention session to within one week after the end of intervention
  computer-based survey for participants to answer questions about isolation
Patient Reported Outcome Measures (PROMIS) Upper Extremity question bank | Within one week before the first intervention session to within one week after the end of intervention
  computer-based survey for participants to answer questions about hand and arm function
Change in size of motor evoked potential in the brain | Within one week before the first intervention session to within one week after the end of intervention
  Using single pulse transcranial magnetic stimulation, we will measure the amount of energy required to evoke a leg muscle movement from a stimulus delivered to the head
Manual Ability Classification System | Within one week before the first intervention session to within one week after the end of intervention
  A categorical measure of how well a participant can move their hands
Jebsen-Taylor Test of Hand Function | Within one week before the first intervention session to within one week after the end of intervention
  A timed test that measures how quickly the participant can move checkers, cans, and small objects

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Friel, PhD, Principal Investigator — Burke Neurological Institute
Locations (1):
- Burke Neurological Institute, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We will email deidentified datasets to other researchers upon request. When we publish our results, we will mention in the paper(s) that the dataset is fully available via email.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available as soon as the findings are published, and will be available indefinitely.
Access Criteria: We will provide data to researchers who have experience with operant conditioning data analyses.

REFERENCES:
- [Background] Thompson AK, Chen XY, Wolpaw JR. Soleus H-reflex operant conditioning changes the H-reflex recruitment curve. Muscle Nerve. 2013 Apr;47(4):539-44. doi: 10.1002/mus.23620. Epub 2012 Dec 21. PMID 23281107
- [Background] Mrachacz-Kersting N, Kersting UG, de Brito Silva P, Makihara Y, Arendt-Nielsen L, Sinkjaer T, Thompson AK. Acquisition of a simple motor skill: task-dependent adaptation and long-term changes in the human soleus stretch reflex. J Neurophysiol. 2019 Jul 1;122(1):435-446. doi: 10.1152/jn.00211.2019. Epub 2019 Jun 5. PMID 31166816